CLINICAL TRIAL: NCT00777257
Title: Immunogenicity and Safety of Meningococcal (Groups A, C, Y, and W-135) Diphtheria Toxoid Conjugate Vaccine (Menactra®) in Adolescents in the US When Administered Concomitantly With Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Tdap Vaccine)
Brief Title: Study of Menactra® in US Adolescents When Administered Concomitantly With Tdap Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTA21
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2009-12-31 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Meningitis; Meningococcemia; Pertussis; Tetanus; Diphtheria
Keywords: Meningitis; Meningococcemia; Pertussis; Neisseria meningitidis; Tetanus; Diphtheria
MeSH Terms: conditions — Meningitis; Meningococcal Infections; Whooping Cough; Tetanus; Diphtheria | interventions — adacel; Meningococcal Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study Group A (Experimental): Tdap vaccine + placebo concomitantly on Day 0; Menactra® vaccine 28 days later
  Interventions: Biological: T dap + Meningococcal Polysaccharide Diphtheria Toxoid Conj.
- Study Group B (Experimental): Tdap vaccine + Menactra® vaccine concomitantly on Day 0; placebo 28 days later
  Interventions: Biological: Tdap + Meningococcal Polysaccharide Diphtheria Toxoid Conj.
- Study Group C (Experimental): Menactra® vaccine + placebo concomitantly on Day 0; Tdap vaccine 28 days later
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conj. + T dap

INTERVENTIONS:
Biological: T dap + Meningococcal Polysaccharide Diphtheria Toxoid Conj. — Day 0: 0.5 mL (T dap)+ Placebo, Intramuscular; Day 28: 0.5 mL (Menactra®) Intramuscular
  Other Names: ADACEL®; Menactra®; Sterile Buffered 0.9% Sodium Chloride
  Arms: Study Group A
Biological: Tdap + Meningococcal Polysaccharide Diphtheria Toxoid Conj. — Day 0: 0.5 mL (T dap) + 0.5 mL (Menactra®) Intramuscular; Day 28: Placebo 0.5 mL Intramuscular
  Other Names: Menactra®; Adacel®; Sterile Buffered 0.9% Sodium Chloride
  Arms: Study Group B
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conj. + T dap — Day 0: 0.5 mL (Menactra®)+0.5 mL Placebo, Intramuscular; Day 28: 0.5 mL (T dap) Intramuscular
  Other Names: Menactra®; Adacel®; Sterile Buffered 0.9% Sodium Chloride
  Arms: Study Group C

SUMMARY:
The purpose of this study was to evaluate the immunogenicity and safety of the concomitant administration of Menactra® vaccine and Tdap vaccine in adolescents aged 11 to 17 years.

Primary Objective:

To determine whether concomitant administration of two vaccines, Tdap and Menactra®, induces antibody responses that are similar to those observed when each vaccine is given separately.

Secondary Objective:

To compare the rates of injection site reactions at the Tdap injection site after Tdap and Menactra® vaccines are administered concomitantly to the corresponding rates of reactions when Tdap vaccine is administered alone.

ELIGIBILITY:
Inclusion Criteria :

* Healthy as determined by medical history and physical examination.
* Aged ≥ 11 to 17 years at the time of study vaccination on Day 0.
* Informed consent form that has been approved by the Institutional Review Board (IRB) signed by the parent or legal guardian.
* Informed assent form that has been approved by the IRB signed by the subject.
* Subject (female) agrees to use measures to prevent pregnancy during the study.

Exclusion Criteria :

* Serious chronic disease (i.e. cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric, etc.).
* Known or suspected impairment of immunologic function.
* Acute medical illness with or without fever within the last 72 hours or an oral temperature ≥ 100.4°F (≥ 38.0°C) at the time of enrolment.
* History of documented invasive meningococcal disease or previous meningococcal vaccination.
* History of documented infection with Bordetella pertussis, Clostridium tetani, or Corynebacterium diphtheriae or vaccination with any tetanus, diphtheria or pertussis vaccine within the previous 5 years.
* Received either immune globulin or other blood products within the last 3 months; or received injected or oral corticosteroids, or other immunomodulator therapy, within 6 weeks of the study vaccines. Individuals on a tapering dose schedule of oral steroids lasting <7 days and individuals (e.g., asthmatics) on a short schedule of oral steroids lasting 3 to 4 days may be included in the trial as long as they have not received more than one course within the last 2 weeks prior to enrolment.
* Received antibiotic therapy within the 72 hours prior to vaccination on Day 0.
* Received any vaccine 28 days prior to the 1st study vaccination or scheduled to receive any vaccination during the course of the study.
* Suspected or known hypersensitivity to either of the two study vaccines or their components.
* Unavailable for the entire study period, or unable to attend the scheduled visits or to comply with the study procedures.
* Enrolled in another clinical trial.
* Diagnosed with any condition, which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* For all females, a positive or equivocal urine pregnancy test at time of study vaccination.
* Nursing mothers.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1345 (Actual)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (20):
- United States (20):
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Boulder, Colorado
  - Marietta, Georgia
  - Woodstock, Georgia
  - Bardstown, Kentucky
  - Baltimore, Maryland
  - Woburn, Massachusetts
  - Albuquerque, New Mexico
  - Syracuse, New York
  - Raleigh, North Carolina
  - Sylva, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Kingsport, Tennessee
  - Spokane, Washington

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 26 April 2005 through 24 June 2005 in 21 Medical centers in the US
Pre-assignment Details: A total of 1345 participants that met the inclusion and exclusion criteria were randomized and vaccinated.
Groups:
- Tdap + Placebo Vaccines Day 0: Participants received Tdap vaccine + placebo concomitantly on Day 0; Menactra® vaccine 28 days later
- Tdap + Menactra® Vaccines Day 0: Participants received Tdap vaccine + Menactra® vaccine concomitantly on Day 0; and Placebo vaccine 28 days later
- Menactra® + Placebo Vaccines Day 0: Participants received Menactra® vaccine + placebo vaccine concomitantly on Day 0; Tdap vaccine 28 days later.
Period: Overall Study
Arm/Group | Tdap + Placebo Vaccines Day 0 | Tdap + Menactra® Vaccines Day 0 | Menactra® + Placebo Vaccines Day 0
Started | 444 | 450 | 451
Completed | 433 | 438 | 442
Not Completed | 11 | 12 | 9
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Lost to Follow-up | 3 | 3 | 2
Not completed — Protocol Violation | 2 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tdap + Placebo Vaccines Day 0 | Tdap + Menactra® Vaccines Day 0 | Menactra® + Placebo Vaccines Day 0 | Total
Number analyzed (Participants) | 444 | 450 | 451 | 1345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 444 | 450 | 451 | 1345.0
  Between 18 and 65 years | 0 | 0 | 0 | 0.0
  >=65 years | 0 | 0 | 0 | 0.0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.0 (1.87) | 13.0 (1.93) | 13.3 (2.05) | 13.1 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 193 | 186 | 599.0
  Male | 224 | 257 | 265 | 746.0
Region of Enrollment [Number; unit: participants]
  United States | 444 | 450 | 451 | 1345.0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 4-fold Rise in Meningococcal Antibody Titer From Baseline (Day 0) to Day 28 Post-vaccination With Menactra® Vaccine.
Time Frame: Day 0 to Day 28 post-vaccination
Population: Serum bactericidal activity using baby rabbit complement (SBA-BR) titers for each meningococcal serogroup was evaluated in the per-protocol population
Measure: Number; unit: Percentage of participants
Arm/Group | Tdap + Placebo Vaccines Day 0 | Tdap + Menactra® Vaccines Day 0 | Menactra® + Placebo Vaccines Day 0
Number analyzed (Participants) | 376 | 382 | 382
Percentage of participants
  Meningococcal Serogroup A | 92 | 94 | 93
  Meningococcal Serogroup C | 80 | 84 | 87
  Meningococcal Serogroup Y | 79 | 87 | 87
  Meningococcal Serogroup W-135 | 94 | 96 | 96

2. Primary Outcome: Geometric Mean Concentrations (GMCs) of Diphtheria and Tetanus Antibodies at Baseline and on Day 28 Post-vaccination With Tdap Vaccine.
Time Frame: Day 0 and Day 28 post-vaccination
Population: Geometric mean concentration for each vaccine antigen was evaluated in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Tdap + Placebo Vaccines Day 0 | Tdap + Menactra® Vaccines Day 0 | Menactra® + Placebo Vaccines Day 0
Number analyzed (Participants) | 377 | 384 | 383
IU/mL
  Diphtheria toxoid - Day 0 | 0.2 [0.2 to 0.3] | 0.3 [0.3 to 0.3] | 56.2 [48.9 to 64.6]
  Diphtheria toxoid - Day 28 | 7.9 [7.0 to 8.8] | 49.8 [43.8 to 56.7] | 38.2 [33.3 to 43.9]
  Tetanus toxoid - Day 0 | 0.9 [0.8 to 0.9] | 0.8 [0.8 to 0.9] | 1.0 [0.9 to 1.1]
  Tetanus toxoid - Day 28 | 22.8 [21.0 to 24.7] | 16.4 [15.2 to 17.5] | 21.1 [19.6 to 22.7]

3. Secondary Outcome: Percentage of Participants Reporting Solicited Injections Site and Systemic Reactions Following Concomitant Administration of Tdap With Placebo; Menactra® With Tdap; and Menactra® With Placebo, Respectively.
Description: Solicited injection sites reactions: Erythema, swelling, and pain. Solicited systemic reactions: Fever (temperature), headache, malaise, and myalgia.
Time Frame: 0 to 7 days post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants intend-to-treat population
Measure: Number; unit: Percentage of participants
Arm/Group | Tdap + Placebo Vaccines Day 0 | Tdap + Menactra® Vaccines Day 0 | Menactra® + Placebo Vaccines Day 0
Number analyzed (Participants) | 444 | 450 | 451
Percentage of participants
  Any Solicited Injection Site Reaction-Tdap, Dose 1 | 87 | 84 | 0
  Grade 3 Solicited Inj. Site Reaction-Tdap, Dose 1 | 10 | 9 | 0
  Any Erythyma (Dose 1) | 25 | 30 | 0
  Grade 3 Erythema (≥ 2 inches, Dose 1) | 4 | 3 | 0
  Any swelling (Dose 1) | 26 | 24 | 0
  Grade 3 swelling (≥ 2 inches, Dose 1) | 5 | 5 | 0
  Any Pain (Dose 1) | 85 | 81 | 0
  Grade 3 Pain (Incapacitating, Dose 1) | 4 | 4 | 0
  Any Solicited Inj. Site Reaction-Menactra, Dose 1 | 0 | 57 | 58
  Grd 3 Solicited Inj Site Reaction-Menactra, Dose 1 | 0 | 4 | 4
  Any Erythyma (Dose 1) | 0 | 19 | 16
  Grade 3 Erythema (≥ 2 inches, Dose 1) | 0 | 2 | 2
  Any swelling (Dose 1) | 0 | 14 | 15
  Grade 3 swelling (≥ 2 inches, Dose 1) | 0 | 2 | 2
  Any Pain (Dose 1) | 0 | 52 | 52
  Grade 3 Pain (Incapacitating, Dose 1) | 0 | 1 | 1
  Any Solicited Inj. Site Reaction-Placebo, Dose 1 | 38 | 0 | 35
  Grd 3 Solicited Inj. Site Reaction-Placebo, Dose 1 | 1 | 0 | 1
  Any Erythyma (Dose 1) | 11 | 0 | 11
  Grade 3 Erythema (≥ 2 inches, Dose 1) | 1 | 0 | 0
  Any swelling (Dose 1) | 11 | 0 | 9
  Grade 3 swelling (≥ 2 inches, Dose 1) | 1 | 0 | 0
  Any Pain (Dose 1) | 33 | 0 | 30
  Grade 3 Pain (Incapacitating, Dose 1) | 0 | 0 | 1
  Any Solicited Injection Site Reaction (Dose 2) | 56 | 24 | 68
  Grade 3 Solicited Inj. Site Reaction (Dose 2) | 4 | 8 | 6
  Any Erythyma (Dose 2) | 13 | 8 | 14
  Grade 3 Erythema (≥ 2 inches, Dose 2) | 2 | 1 | 1
  Any swelling (Dose 2) | 11 | 6 | 14
  Grade 3 swelling (≥ 2 inches, Dose 2) | 2 | 0 | 1
  Any Pain (Dose 2) | 51 | 20 | 65
  Grade 3 Pain (Incapacitating, Dose 2) | 2 | 1 | 5
  Any Solicited Systemic Reaction (Dose 1) | 74 | 69 | 61
  Grade 3 Solicited Systemic Reaction (Dose 1) | 5 | 7 | 3
  Any Fever (Dose 1) | 2 | 4 | 2
  Grade 3 Fever (≥ 40.0 °C, Dose 1) | 0 | 0 | 0
  Any Headache (Dose 1) | 37 | 38 | 37
  Grd 3 Headache (prevents daily activities, Dose 1) | 2 | 4 | 1
  Any Malaise (Dose 1) | 30 | 30 | 25
  Grd 3 Malaise (prevents daily activities, Dose 1) | 3 | 4 | 1
  Any Myalgia (Dose 1) | 60 | 54 | 41
  Grd 3 Myalgia (prevents daily activities, Dose 1) | 2 | 2 | 2
  Any Solicited Systemic Reaction (Dose 2) | 48 | 33 | 54
  Grade 3 Solicited Systemic Reaction (Dose 2) | 4 | 3 | 6
  Any Fever (Dose 2) | 1 | 1 | 1
  Grade 3 Fever (≥ 40.0 °C, Dose 2) | 0 | 0 | 0
  Any Headache (Dose 2) | 27 | 22 | 26
  Grd 3 Headache (prevents daily activities, Dose 2) | 3 | 2 | 3
  Any Malaise (Dose 2) | 19 | 13 | 20
  Grd 3 Malaise (prevents daily activities, Dose 2) | 3 | 1 | 3
  Any Myalgia (Dose 2) | 29 | 15 | 44
  Grd 3 Myalgia (prevents daily activities, Dose 2) | 1 | 1 | 3

4. Primary Outcome: Geometric Mean Concentrations (GMCs) of Pertussis Antibodies at Baseline and on Day 28 Post-vaccination With Tdap Vaccine.
Time Frame: Day 0 and Day 28 Post-vaccination
Population: Geometric mean concentration for each vaccine antigen was evaluated in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Tdap + Placebo Vaccines Day 0 | Tdap + Menactra® Vaccines Day 0 | Menactra® + Placebo Vaccines Day 0
Number analyzed (Participants) | 377 | 384 | 383
EU/mL
  Pertussis Toxoid - Day 0 | 15.3 [13.3 to 17.5] | 14.0 [12.2 to 16.0] | 20.7 [18.0 to 23.9]
  Pertussis Toxoid - Day 28 | 88.0 [79.8 to 97.1] | 73.4 [67.0 to 80.3] | 107.4 [97.6 to 118.2]
  Filamentous Haemagglutinin - Day 0 | 21.4 [18.9 to 24.3] | 20.0 [17.9 to 22.3] | 28.5 [25.4 to 31.9]
  Filamentous Haemagglutinin - Day 28 | 179.5 [163.2 to 197.6] | 140.2 [128.0 to 153.6] | 245.1 [226.4 to 265.2]
  Pertactin - Day 0 | 9.0 [7.9 to 10.3] | 8.4 [7.4 to 9.5] | 11.9 [10.4 to 13.6]
  Pertactin - Day 28 | 176.5 [156.6 to 199.0] | 130.3 [116.5 to 145.9] | 213.6 [192.8 to 236.6]
  Fimbriae Types 2 and 3 - Day 0 | 13.8 [12.0 to 15.9] | 12.7 [11.1 to 14.6] | 14.2 [12.2 to 16.6]
  Fimbriae Types 2 and 3 - Day 28 | 1133.4 [979.3 to 1311.7] | 699.1 [602.9 to 810.7] | 832.3 [712.0 to 972.8]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 2 months post-dose 1 vaccination
Arm/Group | Tdap + Placebo Vaccines Day 0 | Tdap + Menactra® Vaccines Day 0 | Menactra® + Placebo Vaccines Day 0
Serious Adverse Events (participants affected / at risk) | 2/444 | 1/450 | 1/451
Other Adverse Events (participants affected / at risk) | 0/444 | 0/450 | 0/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tdap + Placebo Vaccines Day 0 (N=444) | Tdap + Menactra® Vaccines Day 0 (N=450) | Menactra® + Placebo Vaccines Day 0 (N=451)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.